CLINICAL TRIAL: NCT06236815
Title: High Confusion: Evaluating Effects of Popular Cannabis Isolates on Driving Performance
Brief Title: High Confusion: Cannabis & Driving
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2022-1124; A523000 (Other: UW Madison); Protocol Version 2/5/2025 (Other: UW Madison)
Record Dates: First submitted 2024-01-16; First posted 2024-02-01 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Impairment, Cognitive; Impairment of Attention; Impairment, Psychomotor
Keywords: cannabis; impairment; tetrahydrocannabinol
MeSH Terms: conditions — Cognitive Dysfunction; Psychomotor Disorders; Marijuana Abuse | interventions — Dronabinol; delta-8-tetrahydrocannabinol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- delta-9-THC (Experimental)
  Interventions: Drug: Delta-9-THC
- delta-8-THC (Experimental)
  Interventions: Drug: Delta-8-THC
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Delta-9-THC — Healthy volunteers will attend three test sessions, at least 14 days apart, in which cognition and driving performance will be assessed following vaporization of (1) Δ9-THC, (2) Δ8-THC, or (3) a placebo. The order of these conditions will be counterbalanced across participants. Serial blood samples will be drawn during each dosing visit and compared with concurrent dried blood spots from a finger stick.
  Arms: delta-9-THC
Drug: Delta-8-THC — Healthy volunteers will attend three test sessions, at least 14 days apart, in which cognition and driving performance will be assessed following vaporization of (1) Δ9-THC, (2) Δ8-THC, or (3) a placebo. The order of these conditions will be counterbalanced across participants. Serial blood samples will be drawn during each dosing visit and compared with concurrent dried blood spots from a finger stick.
  Arms: delta-8-THC
Drug: Placebo — Healthy volunteers will attend three test sessions, at least 14 days apart, in which cognition and driving performance will be assessed following vaporization of (1) Δ9-THC, (2) Δ8-THC, or (3) a placebo. The order of these conditions will be counterbalanced across participants. Serial blood samples will be drawn during each dosing visit and compared with concurrent dried blood spots from a finger stick.
  Arms: Placebo

SUMMARY:
This study is being done to assess the feasibility of administrating Δ9-THC and Δ8-THC isolates and simultaneously adopting several data harmonization measures to generate uniquely translatable data. This project aims to (1) evaluate the feasibility and acceptability of administering ∆9-THC and Δ8-THC isolates using standardized cannabis dosing units to quantify ∆9-THC and Δ8-THC pharmacokinetics; and (2) evaluate the feasibility and acceptability of adopting standardized impairment detection methods and driving performance definitions and measures on quantifying ∆9-THC and Δ8-THC driving impairment compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, no older than 49 years of age
* Recent cannabis use (within past two years)
* Good mental health as determined by self-reported responses to the Psychopathology Screener
* Absence of any major medical, cardiovascular, endocrine, and neurological condition as determined by self-reported responses to the Medical History Screener
* In possession of a valid drivers' license with at least two years of driving experience
* English-speaking (able to provide consent and complete questionnaires)
* Written Informed Consent

Exclusion Criteria:

* Any serious prior adverse response to cannabis
* History of or current substance use disorder as determined by self-reported responses to the Internalizing, Externalizing, and Substance Use Disorder Screener
* Pregnancy or lactation (pregnancy test, if needed)
* Use of medications that may impact driving ability (e.g., mood stabilizers, sedatives)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Quantify analyte concentrations | 9 months
  Quantify delta-9-THC, delta-8-THC, and their primary metabolites in whole blood, plasma, oral fluid, and dried blood spots at several time points before and after acute study drug administration.
Quantify impairing effects of cannabinoids | 9 months
  Quantify the impairing effects of delta-9-THC and delta-8-THC by measuring the standard deviation of lateral position within the driving simulation and by completing a drug recognition expert field sobriety test for signs of impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Barkholtz, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No